CLINICAL TRIAL: NCT03909321
Title: Effect of Recreational Beach Tennis on Ambulatory Blood Pressure and Physical Fitness in Hypertensive Individuals (BAH Study)
Brief Title: Beach Tennis And Hypertension Study 2
Acronym: BAH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Collaborators: Federal University of Rio Grande do Sul (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 96487118000005327b
Record Dates: First submitted 2019-04-08; First posted 2019-04-10 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Hypertension
Keywords: Exercise; Beach Tennis; Sport training; Ambulatory blood pressure monitoring
MeSH Terms: conditions — Hypertension; Motor Activity

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): The Control group will not be submitted to intervention and will be instructed not to engage in any kind of structured physical exercise training and to keep the life activities identified at baseline.
- Beach tennis training group (Experimental): The Beach Tennis (BT) group will perform two sessions per week of the Beach Tennis training. This intervention will last 12 weeks.
  Interventions: Behavioral: Beach tennis training group

INTERVENTIONS:
Behavioral: Beach tennis training group — Beach Tennis Training Group (BTG) will perform two sessions of 40-60 min of beach tennis during 12 weeks. BT sessions will be composed by a warm up of 5-10 min of BT technical exercises (i.e., serve, volley, forehand and backhand exercises) followed by 3 BT small games of 10-15 min each.
  Arms: Beach tennis training group

SUMMARY:
No studies have investigated the chronic effects of team sports on 24 h ambulatory blood pressure and have assessed the effects of a beach tennis intervention in cardiovascular profile and physical fitness. Based on that, the investigators designed this parallel randomized controlled trial to evaluate the effect of beach tennis training on 24 h ambulatory blood pressure and different physical fitness parameters in individuals with hypertension. The difference between the intervention arms in mean change from baseline in 24 h, daytime and nighttime systolic and diastolic ambulatory blood pressure at 12-weeks is the primary outcome; secondary outcomes are the difference between mean change in office blood pressure as well as cardiorespiratory fitness, muscular strength and power. The investigators anticipate that 12 weeks of beach tennis training will reduce blood pressure when compared to a non-exercising control group. Additionally, our recreational beach tennis intervention will improve all physical fitness components in comparison to the baseline values.

DETAILED DESCRIPTION:
This is a single-center, two-arms, parallel randomized controlled trial with concealed allocation, blinded measurers, with 12 weeks of follow-up analyzed using an intention-to-treat approach.

Participants will be randomly allocated to the beach tennis training intervention (BTT) or to the control group (Con), which will not be submitted to intervention and will be instructed not to engage in any kind of structured physical exercise training and to keep the life activities identified at baseline. The International Physical Activity Questionnaire (IPAQ) will be applied before and after the intervention in order to assess the level of physical activity.

In BTT, supervised beach tennis sessions will be performed two times per week. Each session will be composed of an initial period of 10 min of warm up and technical exercises (i.e., serve, volley, forehand and backhand). After that, 3 games of 10-15 min each (weeks 1-4: 3 × 10 min; weeks 5-8: 3 × 12 min; and weeks 9-12: 3 × 15 min) with an interval of 2 min between each game will be played in pairs (i.e., 2 versus 2). In case of less than 4 participants are able to play at the same time, the games can also be played individually (i.e., 1 versus1). In Con, participants will be advised to not change their daily usual activities and to not participate in any structured physical exercise program during this period.

ELIGIBILITY:
Inclusion Criteria:

* Office blood pressure between 130-179 and 80-110 mmHg for systolic and diastolic blood pressure, respectively;
* Non-engaged in structured exercise programs in the last 3 months before the beginning of this study;
* Able to perform the proposed exercises.

Exclusion Criteria:

* Underlying cardiovascular disease in the last 24 months such as acute myocardial infarction, angina, stroke or heart failure;
* Diseases that reduce life expectancy;
* Smokers;
* BMI >39.9 kg/m²;
* Diabetic proliferative retinopathy.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2023-02-06 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Ambulatory Blood Pressure | Change from baseline 24-hour systolic blood pressure at 12 weeks
  24h ambulatory blood pressure measured through automatic oscillometric device

SECONDARY OUTCOMES:
Systolic blood pressure | Will be measured during intervention period throughout the first session of weeks 1, 4, 5, 8, 9 and 12.
  Systolic blood pressure in mmHg measured using automatic oscillometric device
Diastolic blood pressure | Will be measured during intervention period throughout the first session of weeks 1, 4, 5, 8, 9 and 12.
  Diastolic blood pressure in mmHg measured using automatic oscillometric device
Cardiorespiratory fitness (Oxygen consumption at peak) | Change from baseline VO2peak at 12 weeks
  Oxygen consumption at peak (VO2peak) as assessed by maximal cardiopulmonary exercise testing
Muscle strength (Test of hand grip strength) | Change from baseline handgrip at 12 weeks
  Performs palmar grip with the greatest possible force
Muscle strength (Chair-stand test) | Change from baseline Chair-stand test at 12 weeks
  The total number of stands executed correctly within 30-s
Muscle strength (Chair-stand test) | Change from baseline Chair-stand test at 12 weeks
  The time to perform the first five stands executed correctly
Power muscle | Change from baseline vertical countermovement jump at 12 weeks
  Vertical countermovement jump tests
Quality of life (WHOQOL-BREF questionnaire) | Change from baseline QoL score at 12 weeks
  The questionnaire contains 26 questions and is divided into four domains (physical, psychological, social and environmental). Responses follow a Likert scale (1 to 5, the higher the score the better the quality of life) and the values of each domain will be expressed in percentage values.
Enjoyment (PACES questionnaire) | Will be measured during intervention period throughout the first session of weeks 1, 4, 5, 8, 9 and 12.
  The scale is composed of 18 items in a bipolar affirmations format (i.e., "amused" versus "not-amused") punctuated in a range from the minimum value "1" to the maximum value "7".

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo Ferrari, PhD, Principal Investigator — Hospital de Clinicas de Porto Alegre
Locations (1):
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Ferrari R, de Oliveira Carpes L, Domingues LB, Jacobsen A, Frank P, Jung N, Santini J, Fuchs SC; BAH Study Group. Effect of recreational beach tennis on ambulatory blood pressure and physical fitness in hypertensive individuals (BAH study): rationale and study protocol. BMC Public Health. 2021 Jan 6;21(1):56. doi: 10.1186/s12889-020-10117-5. PMID 33407276
- [Result] Ferrari R, de Oliveira Carpes L, Betti Domingues L, Mallmann Schneider V, Leal R, Tanaka H, Jung N; The BAH Study Group. Recreational beach tennis training reduces ambulatory blood pressure in adults with hypertension: a randomized clinical trial. J Hypertens. 2024 Dec 1;42(12):2122-2130. doi: 10.1097/HJH.0000000000003850. Epub 2024 Aug 26. PMID 39248124